CLINICAL TRIAL: NCT03121456
Title: 18F-FDG PET Scan and MRI Diffusion : Correlation Study of the Evaluation of the Early Therapeutic Response of Diffuse Large B-cell Lymphoma
Brief Title: 18F-FDG PET Scan and MRI Diffusion.Evaluation of the Early Therapeutic Response of Diffuse Large B-cell Lymphoma
Acronym: LYMPHODTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/12
Record Dates: First submitted 2017-04-12; First posted 2017-04-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDG PET SCAN (Experimental): REALIZATION OF INITIAL 18F-FDG PET SCAN (PRE THERAPEUTIC), THEN BETWEEN CYCLE 2 DAY 10 AND CYCLE 3 DAY 1
  MRI DIFFUSION REALIZATION OF INITIAL MRI DIFFUSION WITHIN 7 DAYS AFTER INITIAL 18F-FDG PET SCAN, THEN WITHIN 7 DAYS AFTER 18F-FDG PET SCAN 1.
  Interventions: Other: 18F-FDG PET SCAN; Other: MRI DIFFUSION

INTERVENTIONS:
Other: 18F-FDG PET SCAN — REALIZATION OF INITIAL 18F-FDG PET SCAN (PRE THERAPEUTIC), THEN BETWEEN CYCLE 2 DAY 10 AND CYCLE 3 DAY 1
Other: MRI DIFFUSION — REALIZATION OF INITIAL MRI DIFFUSION WITHIN 7 DAYS AFTER INITIAL 18F-FDG PET SCAN, THEN WITHIN 7 DAYS AFTER 18F-FDG PET SCAN 1.

SUMMARY:
Open-label, multicenter, uncontrolled and non-randomized study comparing 18F-FDG PET-Scan and diffusion MRI in the assessment of the early therapeutic response of Diffuse Large B-Cell Lymphoma.

DETAILED DESCRIPTION:
High-grade lymphomas are characterized by noisy symptomatology and quick progression kinetics in the absence of treatment. The therapeutic strategy and prognosis of patients depend on the initial staging and evaluation of early therapeutic response. Positron emission tomography injected with labeled fluorodeoxyglucose (18F-FDG PET-CT) is recommended in the initial disease balance; It also has a prognostic value demonstrated in the evaluation of the intermediate and final response of treatment of malignant non-Hodgkin's lymphoma B (LMNH B) to large cells through a qualitative visual analysis using the 5-point scale of Deauville, but also thanks to a quantitative analysis with the measurement of the Delta SUV max. If the 18F-FDG PET-CT is referred to, it is not without constraint, it is notably an examination leading to exposure to ionizing radiation for the patient.

Diffusion MRI (DWI) is a non-irradiating technique based on the evaluation of the diffusion of water molecules allowing indirect qualitative and quantitative analysis of the tumor microstructure, cellularity and integrity of the cell membrane . The tumor is thus detected thanks to its hypercellularity and the mapping of the apparent diffusion coefficient (ADC).

Several recent studies have demonstrated the feasibility and interest of MRI scattering and measurement of CDA in tumor staging and early therapeutic evaluation of high grade lymphomas and more particularly diffuse large B-cell Lyphoma, The latter being characterized by a high nucleo-cytoplasmic cellularity and ratio which makes it possible to obtain a strong signal and low ADC values in diffusion MRI (5) (7) (8) (9) (10) (12) (13) (14). However, there are few studies comparing these two imaging techniques in the therapeutic evaluation of large cell LMNH B (6) (11) (15). The main limitations of the existing studies are their small size and, above all, the accuracy of the methodology for quantifying the measurement of therapeutic response and in particular in terms of quantitative analysis of CDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Diffuse Large B-Cell Lymphoma confirmed histologically
* Patient with a tumor mass defined as measurable according to the RECIST 1.1 criteria,
* Patient requiring a standard first-line chemotherapy treatment (Rituximab -Cyclophosphamide - Hydroxyadriamycin - Oncovin - Prednisone = R-CHOP every 21 days),
* Patient older than 18 years,
* Performance status less than or equal to 2,
* Biological assessment meeting the following criteria: creatinine <150 μmol / l or creatinine clearance> 40 ml / min, total bilirubin <30 μmol / l, transaminases <2.5 x ULN
* Patient of childbearing age must agree to use Means of effective contraception during the treatment period,
* Patient having read the information note and having signed informed consent,
* Patient with Health care insurance available.

Exclusion Criteria:

* History of malignant hemopathy or solid tumor
* History of previous chemotherapy
* Contraindication to one of the examinations studied (Claustrophobia, Pacemaker ...)
* Patient included in another clinical trial for which a period of exclusion is mentioned.
* Patient considered to be a vulnerable person; Vulnerable persons are defined in article L1121-5 to - 8: Pregnant women, women who are pregnant, women who are breastfeeding, Persons deprived of their liberty by a judicial or administrative decision, persons who are hospitalized without consent under Articles L. 3212-1 and L. 3213-1 which do not fall under the provisions of Article L. 1121-8 and persons admitted to a health or social institution for purposes other than research Persons who are the subject of a legal protection measure or are unable to give their consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2024-04-12 (Estimated); Study Completion 2024-04-12 (Estimated)

PRIMARY OUTCOMES:
measurement of the correlation between the Delta SUVmax in PET-TDM (or between the Deauville criteria if the Delta SUVmax is not applicable) and the Delta ADCmax in diffusion MRI. | up to 2 years
  scattering MRI in the assessment of the early therapeutic response of diffuse large cell Lymphoma.

SECONDARY OUTCOMES:
progression free-survival at 2 years | up to 2 years
  Progression-free survival will be assessed between the date of diagnosis and the date of death (any cause) or progression (according to RECIST 1.1) within two years after inclusion.
diagnostic performance of MRI scattering | Up to 4 years
  The diagnostic performance of MRI scattering will be assessed using the following parameters: sensitivity, specificity, positive predictive value (PPV) and negative predictive value (PNP), positive and negative likelihood ratios, area under the ROC as well as the Youden Index. An optimal threshold of the Delta ADCmax will be defined, which will then correspond to a maximum Youden index.
- The degree of inter- and intra-observer association (concordance) of the ADCmax | up to 4 years
  The degree of inter- and intra-observer association (concordance) of the ADCmax will be calculated using the intra-class correlation coefficient (ICC). A representation of Bland and Altman will also be performed in addition to the ICC calculation

CONTACTS AND LOCATIONS:
Overall Officials: Christine LOVERA, Study Director — Centre Antoine Lacassagne
Locations (1):
- Centre antoine-LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided